CLINICAL TRIAL: NCT03072147
Title: Evaluating Teriparatide as a Chondroregenerative Therapy in Human Osteoarthritis
Brief Title: Teriparatide as a Chondroregenerative Therapy in OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Ritchlin (Other)
Collaborators: Eli Lilly and Company (Industry); University of Rochester (Other); Duke University (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor-Investigator, Christopher Ritchlin, Professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Forteo 65996
Record Dates: First submitted 2017-02-21; First posted 2017-03-07 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis; Cartilage Degeneration
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Teriparatide

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, placebo controlled, double blinded study. Interim results will determine if there is a crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Researchers, providers, and subjects will be blinded to treatment group so that outcomes will not be influenced by expectations about the experimental treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1- Treatment (Active Comparator): 20 mcg dosage amounts of teriparatide, in the FDA approved form Forteo, manufactured by Lilly, LLC, are loaded into a 2.4 ml prefilled delivery device (multi injection pen) that administers 28 equal doses as subcutaneous injections in the thigh or abdominal wall. Subjects will inject themselves once a day for 24 weeks.
  Interventions: Drug: Teriparatide
- Group 2- Placebo (Placebo Comparator): Saline placebo is packaged by the manufacturer (Lilly, LLC) in the same 2.4 ml injection pen that is used for teriparatide; it will provide 28 doses of placebo. Subjects will inject themselves once a day for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — 20 mcg of teriparatide injected in thigh or abdomen once a day for 24 weeks.
  Other Names: Group 1; Forteo
  Arms: Group 1- Treatment
Drug: Placebo — 20 mcg of saline injected in thigh or abdomen once a day for 24 weeks.
  Other Names: Group 2
  Arms: Group 2- Placebo

SUMMARY:
The purpose of this study is to evaluate teriparatide (TP) as a chondroregenerative therapy for human knee osteoarthritis (OA). The central hypothesis to be tested is that TP supports structural modification of the joint and improves biomarker, functional and patient-reported measures of knee OA.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo controlled, double blinded, crossover study. The investigators will identify, recruit and enroll 80 subjects with symptomatic, unilateral medial compartment knee OA. Enrolled subjects will be randomized into equal TP (in the FDA approved form, Forteo) or placebo arms of 40 subjects each (includes allowance for a 25% dropout rate with no replacements). All subjects will be treated for 24 weeks, then followed for an additional 24 weeks to assess the durability of any observed effects. The trial incorporates a crossover design, based on interim analysis of the 24 week outcome data after every subject has completed the 24 week treatment period. If positive effects on structural and/or biomarker measures are apparent from the interim analysis, placebo treated subjects will be offered TP (in the FDA approved form, Forteo) and followed for an additional 24 weeks. If the placebo subjects who choose to participate in the crossover treatment have not yet completed the 48 week visit, it will not occur. These subjects will begin the crossover portion 24 week treatment and monitoring period when they receive the TP pens (in the FDA approved form, Forteo).

ELIGIBILITY:
Inclusion Criteria:

1. male or female 40 to 60 years old.
2. radiographic evidence of Kellgren-Lawrence score (K-L score) grade I-II OA in the affected knee
3. unilateral symptomatic knee OA
4. willingness to forgo potential standard of care treatments (hyaluronic acid and cortisol injections) for knee pain for the duration of the study
5. body Mass Index of ≤40
6. normal screening vitamin D levels (≥20 and ≤100 mg/ml)
7. normal screening serum calcium level (8.5- 10.2 mg/dL)
8. a negative screening serum pregnancy test for premenopausal women

Exclusion Criteria:

1. history of primary hyperparathyroidism disease, hypercalcemia, or persistently abnormal intake PTH levels (≥10 or ≤65 pg/ml)
2. history of musculoskeletal malignancy or solid organ carcinoma
3. active renal disease defined by a creatinine clearance of <35 or history of kidney stones within the past year
4. use of anticonvulsant or digoxin therapy
5. inflammatory disease (bowel disease, spondylitis, lupus, fibromyalgia, psoriasis, rheumatoid arthritis, etc)
6. current or past treatment with teriparatide
7. use of immunosuppressants
8. severe claustrophobia, retained eye or skull metal fragments, metal hardware in or around the affected knee or other standard contraindications to MRI (cochlear implants, pacemakers)
9. dementia, cognitive impairment or other factors that referring provider feels would prevent ability to obtain informed consent and/or follow study protocol
10. pregnancy or intent to become pregnant in the two and a half years following enrollment
11. women who are currently breastfeeding
12. Paget's disease
13. osteoporosis diagnosis by DXA in medical history (T-score less than or equal to -2.5)
14. reliance on assistive walking devices (canes, walkers, braces, etc.)
15. participation in concurrent clinical studies involving investigational medications

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Knee MRI | Change from Baseline through study completion (baseline, 24 weeks, 48 weeks), an average of one year.
  Analysis using Regional Cartilage Volume Segmentation

SECONDARY OUTCOMES:
Flexed Knee Radiograph | Change from Baseline through study completion (baseline, 24 weeks, 48 weeks), an average of one year.
  Interpreted using fractal signature analysis.
Urine Biomarker Analysis | Change from Baseline through study completion (baseline, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  Analyzed immediately via enzyme-linked immunosorbent assay (ELISA) to quantify the following biomarker: urinary type II collagen
Serum Biomarker Analysis | Change from Baseline through study completion (baseline, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  Analyzed immediately via enzyme-linked immunosorbent assay (ELISA) to quantify the following biomarker: serum type II collagen degradation neoepitope.
GAITRite | Change from Baseline through study completion (baseline, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  Change in gait pre- and post-treatment analyzed using the GAITRite walking test.
Timed up and go | Change from Baseline through study completion (baseline, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  Change in gait pre- and post-treatment analyzed using the timed-up-and-go (TUG) test.
WOMAC 3.1 | Change from Baseline through study completion (baseline, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC 3.1) measures pre- and post-treatment changes in subjective pain and functionality.
PROMIS Depression | Change from Baseline through study completion (baseline, 4 weeks, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  The Depression scale from the Patient-Reported Outcomes Measurement Information System (PROMIS) measures measures subjective changes in mood, pre- and post-treatment.
PROMIS Pain Interference | Change from Baseline through study completion (baseline, 4 weeks, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  The Pain Interference scale from the Patient-Reported Outcomes Measurement Information System (PROMIS) measures subjective changes in pain distress, pre- and post-treatment.
PROMIS Physical Function | Change from Baseline through study completion (baseline, 4 weeks, 12 weeks, 24 weeks, 48 weeks), an average of one year.
  Physical function scale from the Patient-Reported Outcomes Measurement Information System (PROMIS) measures subjective changes in mobility and activities of daily living, pre- and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zuscik, PhD, Principal Investigator — University of Rochester; Emily Carmody, MD, Principal Investigator — University of Rochester; Christopher Ritchlin, MD, Principal Investigator — University of Rochester
Locations (1):
- URMC Orthopaedics, Clinton Crossings Building D, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No